CLINICAL TRIAL: NCT03010332
Title: An Expanded Access Protocol of ATA230 (Third-Party Donor-Derived Cytomegalovirus-Specific T Cells) for the Treatment of CMV Viremia or Disease in Subjects for Whom There Are No Other Comparable Options
Brief Title: Expanded Access Protocol of ATA230 (Third-Party Donor-Derived CMV-CTLs) for the Treatment of CMV Viremia or Disease
Status: No longer available | Type: Expanded Access
Sponsor: Atara Biotherapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: ATA230-EAP-201
Record Dates: First submitted 2017-01-03; First posted 2017-01-05 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: CMV Viremia; CMV Disease
Keywords: Cytomegalovirus; Cytomegalovirus Viremia; Cytomegalovirus Infection; CMV Infection; Hematopoietic Cell Transplant; Solid Organ Transplant; Human Immunodeficiency Virus; Cytomegalovirus Disease; Hematopoietic Stem Cell Transplant; CMV; CMV syndrome; Cytomegalovirus syndrome; CMV disease; CMV viremia; allogeneic; third-party
MeSH Terms: conditions — Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome

INTERVENTIONS:
Biological: Cytomegalovirus-specific Cytotoxic T Lymphocytes (CMV-CTLs) — ATA230 (third-party donor-derived CMV-CTLs) are cytotoxic T lymphocytes that specifically kill cells presenting CMV protein antigens.
  Other Names: ATA230

SUMMARY:
This is an expanded access protocol designed to provide access of ATA230 to subjects with cytomegalovirus (CMV) viremia or disease, who are intolerant to, or failed, standard antiviral therapy and have no comparable treatment options.

DETAILED DESCRIPTION:
ATA230 (third-party donor-derived CMV-CTLs) are cytotoxic T lymphocytes that specifically kill cells presenting CMV protein antigens.

This is an expanded access protocol designed to provide access of ATA230 to subjects with CMV viremia or disease, who are intolerant to, or failed, standard antiviral therapy and have no comparable treatment options. This study will enroll subjects regardless of the underlying susceptibility to CMV, including allogeneic hematopoietic cell transplant (alloHCT), solid organ transplant (SOT), human immunodeficiency virus (HIV), other immunocompromised states, and immune competent subjects who require therapy. Subjects must have active CMV viremia or disease for ≥ 2 weeks despite treatment with antiviral therapy or must be intolerant to antiviral therapy due to treatment-related toxicity or comorbidities such as renal insufficiency or myelosuppression.

ATA230 will be administered in cycles lasting 5 weeks (35 days). During each cycle, subjects will receive intravenous (IV) ATA230 at a dose of 1×10^6 cells/kg (with an acceptable range of 0.8-1.0×10^6 cells/kg) on Days 1, 8, and 15, followed by observation through Day 35.

ELIGIBILITY:
Inclusion Criteria:

A subject will be considered eligible to participate in the study if the following inclusion criteria are satisfied:

1. Has a clinically documented condition associated with CMV disease (eg, interstitial pneumonia, hepatitis, encephalitis, retinitis, colitis) or microbiological evidence of CMV viremia or tissue invasion with CMV infection (as determined by viral culture or levels of CMV DNA in blood or body fluids)
2. The CMV disease or CMV viremia is characterized by at least one of the following:

   1. CMV disease is persistent or clinically progressing despite ≥ 2 weeks of antiviral therapy
   2. CMV viremia/disease is persistent or increasing (determined by quantitation of blood CMV DNA) despite ≥ 2 weeks of antiviral therapy
   3. A genetic mutation associated with antiviral drug resistance is present
   4. Unable to continue antiviral drugs due to drug-associated toxicity.
3. No other comparable or satisfactory therapies are available for treatment of CMV
4. Not eligible for any other trials supporting development of ATA230
5. For subjects who received an alloHCT, the underlying disease for which the alloHCT was performed is in morphologic remission
6. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 3× the upper limit of normal (ULN) and total bilirubin < 2.5×ULN unless caused by CMV
7. Availability of appropriate ATA230 cell lot (ie, HLA partially-matched and restricted CMV-CTLs)
8. Subject or subject's representative is willing and able to provide written informed consent

Exclusion Criteria:

A subject will not be eligible to participate in the study if any of the following criteria are met:

1. Receiving concomitant investigational therapy (co-enrollment in a non-interventional study or a study for follow-up or sample collection only is permitted)
2. Need for antimetabolite agents (eg, methotrexate), or extracorporeal photopheresis
3. Antithymocyte globulin or similar anti-T cell antibody therapy ≤ 4 weeks prior to the first dose of ATA230 (on Day 1 of Cycle 1)
4. Need for vasopressor or ventilator support
5. Pregnancy, except when ATA230 is clearly needed
6. Female of childbearing potential or male with a female partner of childbearing potential unwilling to use a highly effective method of contraception
7. Inability to comply with study procedures

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Willis Navarro, MD, Study Director — Atara Biotherapeutics